CLINICAL TRIAL: NCT05356793
Title: A Double-Masked, Placebo-Controlled, Randomized, Phase II Clinical Trial To Assess The Efficacy Of SCH1 In The Treatment Of Acute Infectious Conjunctivitis
Brief Title: The Efficacy Of SCH1 In The Treatment Of Acute Infectious Conjunctivitis
Acronym: SCH1TAIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sacsh (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCH-1001
Record Dates: First submitted 2022-04-10; First posted 2022-05-02 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2022-04

CONDITIONS: Acute Infectious Conjunctivitis (Disorder)
Keywords: Conjunctivitis; Eye
MeSH Terms: conditions — Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Active treatment with SCH-1
  Interventions: Drug: SCH-1
- Placebo (Placebo Comparator): Vehicle minus active components
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCH-1 — Novel anti-infective eyedrop
  Arms: Treatment
Drug: Placebo — SCH-1 vehicle minus active components eyedrop
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy of Sasch1, a novel anti-infective eyedrop, in the treatment of acute infectious conjunctivitis.

DETAILED DESCRIPTION:
This is a Phase II single-center, double-masked, placebo controlled, randomized study of SCH1 for the treatment of infectious conjunctivitis. Approximately 30 subjects will be enrolled, who will be randomized in a 1:1 ratio between SCH1and placebo. Subjects will be assessed at day 1, day 3, and day 5 for efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Conjunctivitis (as defined below) within 72 hours of initial ocular symptoms.
* At least 18 years of age.
* Subjects capable of understanding the purpose and risks of the study, and able to give informed consent.
* Conjunctivitis diagnosis defined as presence of the two cardinal signs of acute conjunctivitis- 1) bulbar conjunctival injection and 2) conjunctival discharge/exudates.
* A three-point rating scale (0=absent, 1=mild, 2=moderate, 3=severe) will be employed to grade conjunctival discharge/exudates.
* All patients will require a rating of 1(mild) or greater for conjunctival discharge/exudates.
* Patients will require a rating of 1 (mild) for bulbar conjunctival injection.

Exclusion Criteria:

* Conjunctivitis greater than 72 hours after initial ocular symptoms
* Corneal ulcer, endophthalmitis, or any other confounding infection of the eye
* Patients taking topical anti-inflammatory medications on a chronic basis
* Known steroid glaucoma responders
* Active herpes ocular infection
* Pregnant women
* Known allergy to chlorhexidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-13 (Actual); Study Completion 2022-08-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Clinical Resolution Among Who Received SCH1 or Placebo on Day 5 | Day 5
  Clinical resolution was defined as absence (score=0) of bulbar conjunctival injection and ocular conjunctival discharge in the study eye. Bulbar conjunctival injection was assessed based on 0 (Normal conjunctival vascular pattern) - 3 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from validated bulbar redness (VBR) scale. Ocular conjunctival discharge was assessed based on 0 (No evidence of discharge in conjunctiva) - 3 (Abundant quantity of mucopurulent or purulent discharge) scale. The study eye was defined as an eye with score of at least 1 for both ocular conjunctival discharge and bulbar conjunctival redness at baseline. Data analysis was performed in SCH1 and placebo reporting groups.

CONTACTS AND LOCATIONS:
Overall Officials: David Ritterband, MD, Principal Investigator — Sacsh
Locations (1):
- Jacqueline Dauhajre, MD, Jackson Heights, New York, United States

IPD SHARING:
Plan to Share IPD: No